CLINICAL TRIAL: NCT00265135
Title: A Phase I/II Study of a Chimeric Antibody Against Interleukin-6 (CNTO 328) in Subjects With Metastatic Renal Cell Carcinoma
Brief Title: A Study of CNTO 328 in Subjects With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005278; C0328T01 (Other: Centocor)
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal cell carcinoma; CNTO 328; Infusions; Renal cell cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part 1 (CNTO 328) (Experimental): In Part 1 of the study, 4 intravenous infusions (IV) [injection of a substance into a vein] of CNTO 328 will be administered to patients in 4 dose levels ranging from 1, 3, 6, and 12 mg/kg on days 1, 29, 43, and 57 to determine the maximum tolerated dose for Part 2 of the study.
  Interventions: Drug: CNTO 328
- Part 2 (CNTO 328) (Experimental): In Part 2 of the study, 2 well tolerated dose levels of CNTO 328 from Part 1 of the study will be administered every 3 weeks as 4 IV infusions to patients.
  Interventions: Drug: CNTO 328
- Part 3 (CNTO 328) (Experimental): In Part 3 of the study, CNTO 328 at a dose level of 6 mg/kg will be administered as IV infusion every 2 weeks for at least 6 doses.
  Interventions: Drug: CNTO 328

INTERVENTIONS:
Drug: CNTO 328 — Patients will receive CNTO 328 at dose levels ranging from 1, 3, 6, and 12 mg/kg in Part 1 of the study to determine the maximum tolerated dose for Part 2 of the study. Patients will receive 2 well tolerated dose levels of CNTO 328 from Part 1 of the study every 3 weeks in Part 2 of the study. Patients will receive 6 mg/kg of CNTO 328 every 2 weeks in Part 3 of the study.

SUMMARY:
The purpose of this study is to better understand the safety, tolerability and distribution of CNTO 328 in the bloodstream.

DETAILED DESCRIPTION:
This research study uses a type of drug called anti-IL-6 monoclonal antibody, also known as CNTO 328. CNTO 328 is a new experimental drug. This study is trying to better understand the safety, the tolerability (side effects), and the distribution of the drug in the blood stream. The effects of CNTO 328 in patients with renal cell carcinoma are currently unknown. However, recent data has shown that treatment with another anti-IL-6 monoclonal antibody reduces the symptoms of renal cell carcinoma.

The study is divided in 3 parts. Part 1 is the phase I portion of the study and evaluated the safety of CNTO 328 in subjects with metastatic renal cell carcinoma. Part 2 and 3 will evaluate efficacy and safety of the drug in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis (histologically confirmed, preferably) of metastatic renal cell carcinoma with documented metastases beyond the level of the regional lymphatics (ie, any T, any N, M1 disease)
* Measurable or evaluable disease (Part 1); measurable disease (Part 2 and Part 3)
* Documented disease progression based on objective tumor assessment (Part 2 and Part 3), proven by tumor measurements on 2 computerized tomography scans within 6 months prior to enrollment
* Life expectancy greater than or equal to 6 months at screening
* Serum C-reactive protein (CRP): detectable ( 4 mg/L or more) according to the standard assay of the core laboratory (Part 1 and Part 2); serum CRP detectable to 30 mg/L or more (Part 3)

Exclusion Criteria:

* Received any investigational drug within 30 days, whichever is longer
* History of receiving murine or chimeric proteins or human/murine recombination products (such as BE8 and other anti-IL-6 monoclonal antibodies)
* Serious concurrent illness or significant cardiac disease characterized by significant ischemic coronary disease or congestive heart failure
* Chronic infection, prior history of recurrent infection, or clinically important active infection
* Presence of a transplanted solid organ (with the exception of a corneal transplant more than 3 months prior to screening) or having received an allogeneic bone marrow transplant or peripheral blood stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2003-08; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Number of Patients With Dose-limiting Toxicity as a Measure of Safety (Parts 1 and 3) | Up to 6 weeks after the last dose
Number of Patients With Tumor Response (Parts 2 and 3) | Up to Week 11
  Tumor response will be evaluated as sum of complete response (CR) and partial response (PR). CR is disappearance of all measurable and evaluable disease. No new lesions. No evidence of non evaluable disease. PR is 50% or more decrease from baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions.
Serum Concentration of CNTO 328 (Parts 1, 2, and 3) | Pre dose, up to 6 weeks after the last dose
Number of Participants With Adverse Events (Parts 1, 2, and 3) | Up to 6 weeks after the last dose
Change From Baseline in C-reactive Protein (Part 1) | Within 2 weeks before first dose, pre dose, post dose (6 weeks after the last dose)
Change From Baseline in Interleukin-6 levels (Part 1) | Within 2 weeks before first dose, pre dose, post dose (6 weeks after the last dose)

SECONDARY OUTCOMES:
Serum Antibodies to CNTO 328 (Parts 1, 2, and 3) | Up to 6 weeks after the last dose
  Serum levels of antibodies to CNTO 328 will be used to evaluate potential immunogenicity.
Number of Patients With Clinical Benefit (Parts 1, 2, and 3) | Up to 6 weeks after the last dose
  Clinical benefit will include assessment of pain (measured using Brief Pain Inventory which includes 4 items assessing pain intensity (pain intensity subscales) and 7 items assessing how much pain has interfered with daily activities (pain interference subscales). The pain intensity score is assessed with 4 questions rated on 11-point numerical rating scale (NRS) ranging from "0 = no pain" to "10 = higher severity of pain". The pain interference score is assessed with 7 questions rated on 11-point numerical rating scale (NRS) ranging from "0 = does not interfere" to "10 = completely interferes". Higher scores indicate worsening), functional impairment (assessed using Karnofsky performance status which quantifies patient's well-being and activities of daily life), weight change (assessed by change in body weight).
Time to disease progression (Parts 2 and 3) | Up to 6 weeks after the last dose
  Disease progression is defines as greater than or equal to 25% increase in the sum of products of measurable lesions over the smallest sum observed (over baseline if no decrease) using the same techniques as baseline, or clear worsening of any evaluable disease, or reappearance of any lesion which had disappeared, or appearance of any new lesion, or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Duration of Tumor Response (Parts 2 and 3) | Screening (3 weeks prior to first dose), Week 7, Week 11, and 6 weeks after the last dose
  Duration of tumor response is defined as sum of complete response which is complete disappearance of all measurable and evaluable disease. No new lesions. No evidence of nonevaluable disease and partial response which is 50% or more decrease from baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions.
Number of Patients With an Overall Tumor Response (Parts 2 and 3) | Screening (3 weeks prior to first dose), Week 7, Week 11, and 6 weeks after the last dose
  Overall tumor response is defined as sum of overall CR which is 2 or more objective responses of CR (complete disappearance of all measurable and evaluable disease.) documented for a minimum of 4 weeks apart, overall PR which is 2 or more objective responses of PR (50% or more decrease from baseline in the sum of products of perpendicular diameters of all measurable lesions.) or better documented for a minimum of 4 weeks apart, and overall stable disease which is at least 1 objective response of SD (radiologic assessments have been evaluated and does not qualify for CR, PR, or progressive disease) at least 3 weeks after baseline.
Change From Baseline in Quality of Life Measured Using Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue questionnaire (Parts 1, 2, and 3) | Within 2 weeks before dose, prior to first dose, Days 29, 43, 57, and 71, and 6 weeks after the last dose
  FACIT - Fatigue scale is a questionnaire to assess fatigue. It is a 13-item questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. Responded to each area are scored from 0 (not at all) to 4 (very much). Higher scores indicate worsening.
Change From Baseline in C-reactive Protein (Parts 2 and 3) | Within 2 weeks before first dose, pre dose, post dose (6 weeks after the last dose)
Change From Baseline in Interleukin-6 levels (Parts 2 and 3) | Within 2 weeks before first dose, pre dose, post dose (6 weeks after the last dose)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (14):
- Czechia (2):
  - Brno
  - Hradec nad Svitavou
- France (5):
  - Caen
  - Lyon
  - Montpellier
  - Montpellier Cedex 5 N/A
  - Villejuif
- Netherlands (3):
  - Groningen
  - Nijmegen
  - Rotterdam
- United Kingdom (4):
  - Birmingham
  - Leeds
  - Manchester
  - Plymouth

REFERENCES:
- See also: A Phase 1/2 Study of a Chimeric Antibody Against Interleukin-6 (CNTO 328) in Subjects with Metastatic Renal Cell Carcinoma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=159&filename=CR005278_CSR.pdf